CLINICAL TRIAL: NCT00795964
Title: Influence of Tidal Volume on Postoperative Pulmonary Function
Acronym: tidalvolume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Dr. med. Tanja A. Meyer-Treschan, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Intraoperative tidalvolume-25
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Pulmonary Function
Keywords: tidal volume; predicted body weight; lung function; respiratory outcome; Respiratory Function Tests; surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): intraoperative mechanical ventilation with 6 ml/kg predicted body weight
  Interventions: Other: Randomized application of intraoperative tidal volume
- 2 (Active Comparator): intraoperative mechanical ventilation with 12 ml/kg predicted body weight
  Interventions: Other: Randomized application of intraoperative tidal volume

INTERVENTIONS:
Other: Randomized application of intraoperative tidal volume — intraoperative mechanical ventilation with 6 ml/kg predicted body weight
  Other Names: Respiratory management
  Arms: 1
Other: Randomized application of intraoperative tidal volume — intraoperative mechanical ventilation with 12 ml/kg predicted body weight
  Other Names: Respiratory management
  Arms: 2

SUMMARY:
Lung function impairment is common after abdominal surgery. Few preventive strategies exist against postoperative lung function impairment. A new potential preventive strategy against postoperative lung function impairment comes from research on critically ill patients with severe respiratory failure. In this field research has long focused on influence of breathing volume (= tidal volume) during mechanical ventilation on outcome. It has been shown, that low tidal volumes improve patients outcomes as compared to (conventional) high tidal volumes. Therefore, we propose a patient and investigator blinded randomised trial to test the hypotheses that intraoperative mechanical ventilation with low tidal volumes as compared to high tidal volumes reduces postoperative lung function impairment in high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age ≥ 50 years and ASA classification ≥ II
* elective upper abdominal surgery of at least 3 hours duration
* general anaesthesia plus epidural anaesthesia.

Exclusion Criteria:

* < 18 years of age
* impaired mental state
* unwillingness to participate
* pregnancy
* duration of surgery < 3 hours
* ASA physical status ≥ IV
* increased intracranial pressure
* neuromuscular disease that impairs spontaneous breathing

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Lung function as assessed by spirometry | 1 year

SECONDARY OUTCOMES:
lung function as assessed by blood gas analysis | 1 year
time till hospital discharge | 1 year
postoperative organ dysfunction | 1 year
postoperative chest x-rays | 1 year
time till mobilisation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tanja A Meyer-Treschan, MD, Principal Investigator — Department of Anesthesiology at Duesseldorf University Hospital
Locations (1):
- Department of Anesthesiology, Düsseldorf, Germany